CLINICAL TRIAL: NCT06253312
Title: Comparison of Open Surgery, Hybrid and Endovascular Repair for Complex TASC C/D Aortoiliac Lesions
Brief Title: Treatment of TASC C and D Aortoiliac Lesions
Status: Recruiting | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: University of Belgrade (Other); University of Trieste (Other); Centro Hospitalar De São João, E.P.E. (Other); Clinical Center Nis, University of Nis (Unknown); Clinical Center Novi Sad, University of Novi Sad (Unknown); Institute for Cardiovascular Diseases Dedinje (Other)
Responsible Party: Principal Investigator, Petar Zlatanovic, Principal investigator, Clinical Centre of Serbia
Other Study IDs: Complex aortoiliac lesions
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease; Aortoiliac Occlusive Disease; Leriche Syndrome; Peripheral Vascular Disease
Keywords: peripheral arterial disease; aortoiliac disease; TASC C,D; open surgery; hybrid repair; endovascular repair; atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Leriche Syndrome; Peripheral Vascular Diseases; Atherosclerosis | interventions — Conversion to Open Surgery; Axillofemoral Bypass Grafting; Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open surgery: Patients with complex TASC C and D aortoiliac occlusive disease undergoing open surgery: aortobifemoral bypass, crossover bypass, axillobifemoral bypass, aortoiliac endarterectomy, iliofemoral bypass
  Interventions: Procedure: Open surgery
- Hybrid repair: Patients with complex TASC C and D aortoiliac occlusive disease undergoing simultaneous open surgical femoral artery reconstruction (endarterectomy, bypass, profundoplasty) and stenting of the iliac axis
  Interventions: Procedure: Hybrid repair
- Endovascular repair: Patients with complex TASC C and D aortoiliac occlusive disease undergoing total endovascular repair using different material: bare metal stents (self and balloon expandable), stent-grafts (self and balloon expandable), covered endovascular reconstruction of aortic bifurcation (CERAB), simple plain old balloon angioplasty (POBA)
  Interventions: Procedure: Endovascular repair

INTERVENTIONS:
Procedure: Open surgery — Patients with complex TASC C and D aortoiliac occlusive disease undergoing open surgery: aortobifemoral bypass, crossover bypass, axillobifemoral bypass, aortoiliac endarterectomy, iliofemoral bypass
  Other Names: Aortobifemoral bypass; Crossover bypass; Axillobifemoral bypass; Aortoiliac endarterectomy; Iliofemoral bypass
  Groups: Open surgery
Procedure: Hybrid repair — Patients with complex TASC C and D aortoiliac occlusive disease undergoing simultaneous open surgical femoral artery reconstruction (endarterectomy, bypass, profundoplasty) and stenting of the iliac axis
  Other Names: Iliac stenting; Femoral endarterectomy
  Groups: Hybrid repair
Procedure: Endovascular repair — Patients with complex TASC C and D aortoiliac occlusive disease undergoing total endovascular repair using different material: bare metal stents (self and balloon expandable), stent-grafts (self and balloon expandable), covered endovascular reconstruction of aortic bifurcation (CERAB), simple plain old balloon angioplasty (POBA)
  Other Names: Bare metal stenting; Covered stent; Plain old balloon angioplasty
  Groups: Endovascular repair

SUMMARY:
Background:

The treatment of patients with complex aortoiliac disease (AID), classified as Trans-Atlantic Inter-Society consensus II (TASC) class C and D, presents a dilemma for vascular surgeons. Current guidelines recommend either open surgical reconstruction (OR), hybrid repair (HR) combining iliac stenting with femoral endarterectomy, or total endovascular repair (ER). While traditional OR with aortobifemoral bypass (ABF) is associated with excellent long term patency results, it is associated with significant perioperative morbidity with some studies citing mortality rates of up to 4-8%. The advancement of endovascular techniques has led to many trials suggesting that endovascular management of TASC II C and D lesions is a potential alternative treatment to open strategies mainly in the subset of patients with high surgical risk, given the substantially less perioperative morbidity and mortality compared to OR.

Aim:

The aim of this trial is to evaluate the short, mid-, and long-term results of open repair, hybrid and endovascular repair in the treatment patients with complex, TASC C and D, aortoiliac lesions.

Methodology:

This is a retrospective cohort study planning to include vascular surgery centers from the following countries: Italy, Portugal, Spain, and Serbia. Data will be collected on demographics, baseline comorbidities, anatomy and morphology of the aortoiliac and femoral bifurcation disease, intraoperative, postoperative, and follow-up data. Propensity score analysis will be performed by matching open repair patients in all three groups (open, hybrid, and endovascular repair) controlling for demographics, baseline comorbidities, anatomical and morphological data.

Endpoints:

Primary endpoints are all-cause mortality and the major adverse limb events (major amputation - below and above the knee, new onset acute limb ischaemia, reintervention of the treated arterial segment). The secondary endpoints are the 30-day complications and primary patency.

DETAILED DESCRIPTION:
Background:

The treatment of patients with complex aortoiliac disease (AID), classified as Trans-Atlantic Inter-Society consensus II (TASC) class C and D, presents a dilemma for vascular surgeons. Current guidelines recommend either open surgical reconstruction (OR), hybrid repair (HR) combining iliac stenting with femoral endarterectomy, or total endovascular repair (ER). While traditional OR with aortobifemoral bypass (ABF) is associated with excellent long term patency results (85%-90% at five years and 75%-80% at ten years), it is associated with significant perioperative morbidity with some studies citing mortality rates of up to 4-8%. HR has evolved as an attractive minimally invasive alternative to OR, especially if the disease extends to the femoral bifurcation, with the potential advantages of lower perioperative morbidity and a shorter hospital stay. On the other hand, ER offers an attractive alternative with durable results (five-year primary and secondary patency rates ranging from 60% to 86% and 80% to 98%, respectively), especially in less extensive AID. When combined with low perioperative morbidity it makes ER generally preferable for patients with more severe co-morbid conditions. Thus, surgical approaches for extensive AID have changed considerably over the last years, primarily due to increased ER. The advancement of endovascular techniques has led to many trials suggesting that endovascular management of TASC II C and D lesions is a potential alternative treatment to open strategies mainly in the subset of patients with high surgical risk, given the substantially less perioperative morbidity and mortality compared to OR. However, currently, there are no randomized control trials nor large observational trials comparing these treatment option for complex (TASC C and D) aortoiliac lesions. Vascular surgeons are therefore left with a paucity of data to guide decision-making.

Sample size:

To ensure sufficient statistical power to answer hypothetical questions, approximately 900 subjects will be entered into the database. Major adverse limb event rate is the primary endpoint being used to calculate the sample size. Assuming a difference in terms of MALE, 243 patients would be required in each arm to achieve a statistical power of 85% at p=0.05. With three arms (endovascular versus open), assuming a 20% rate of missing data, a total N of 875 patients is required.

Research Design

This is a retrospective study including patients with peripheral arterial disease (all Rutherford stages) treated for TASC C/D aortoiliac lesion from January 1st 2015 until January 1st 2022 in four European countries: Italy, Portugal, Spain, and Serbia.

Procedures Involved:

The study does not involve any patient contact and will not impact the care that patients receive. Data regarding the patients will be compiled and analyzed to accomplish the proposed study objectives. Data collection will include demographic information, patient-related factors, and comorbidities, diagnostic imaging information (describing the morphology of aortoiliac segment and femoral bifurcation), laboratory data, surgical procedure information, complications of the surgery, short- and long-term clinical outcomes.

Multi-Institutional research:

After the data has been collected at a participating institution, the data will be transmitted to online database which will be available only to a central analytic center located at the Clinic for Vascular and Endovascular Surgery/University Clinical Center of Serbia/Medical Faculty, University of Belgrade.

Risks to Subjects:

As this is a retrospective observational study with prospective character, there is no potential for physical risks to subjects. There is a minimal risk of breach of confidentiality that could occur when patient information is collected and analyzed for the proposed study. However, appropriate measures will be taken to minimize the risk as much as possible. All information recorded will be de-identified. This study will abide by all regulations related to protecting human subjects and protected health information.

Potential Benefits to Subjects:

There is no direct benefit to the subjects. However, future patients treated with complex TASC C/D aortoiliac lesions where every treatment option is feasible may benefit from improved care as a result of this study.

Statistics and Data Analysis:

Continuous variables will be described using the median and interquartile range or mean and standard deviation. Categorical variables will be described using frequencies and percentages. Group comparisons will be performed by using the Student t-test or Mann-Whitney U test, as appropriate. Categorical data will be expressed as percentages and were compared using the chi-square test or Fisher exact test. Propensity score analysis will be performed by matching endovascular to OR, HR, and ER group in a 1:1:1 ratio controlling for demographics, baseline comorbidities, and imagining parameters. Differences will be considered statistically significant at p < 0.05. The cumulative incidences of all-cause mortality, MALE, and primary patency rates will be estimated using the Kaplan-Meier method. Differences between curves will be tested using the log-rank test. Binary outcomes will be evaluated first by univariable methods, with results reported as odds ratio (OR) with 95% confidence intervals (CI). A multiple logistic regression model will be built including significant co-variables and confounders based on univariable screen (p < 0.1) or because of clinical significance. A multivariable Cox proportional hazard will be used to assess independent predictors for long-term outcomes with results reported as hazard ratio (HR) with 95% CI. Covariables for these models will be selected based on previously described risk factors and the univariable screen of all available potential confounders. Analyses will be done with SPSS software, version 28.0 (SPSS, Chicago, ILLINOIS, USA).

Conflict of Interest:

The investigators have no conflict of interest to report.

Funding Source:

There are no plans to apply for grants or additional funding. No funding is required for the completion of this study.

Publication Plan:

All research personnel included in this project will be eligible for authorship in any resulting abstracts and publications in accordance with the qualifications outlined by the International Committee of Medical Journal Editors. The order of authors will be determined prior to manuscript development and depend on each individual's contribution to the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients (over 18 years of age) with a history of atherosclerotic peripheral arterial disease treated between 1st January 2015 and 1st January 2022
* All management strategies will be included (endovascular, hybrid, and open)

Exclusion Criteria:

* Patients who are pregnant
* Patients who are under 18 years of age
* Patients who have acute limb ischemia or acute on chronic ischemia
* Non-atherosclerotic origin of disease: cyclist disease, trauma, dissection
* Patients who were treated in conservative manner
* Patients who underwent primary major amputation
* Patients with limited life expectancy (less than 2 years)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with peripheral arterial disease according to the Rutherford classification system (with claudications and chronic-limb threatening ischemia) undergoing one of the three available treatment option:
  * Open surgery (aortobifemoral bypass, aortoiliac endarterectomy, iliacofemoral bypass, crossover bypass, axillobifemoral bypass)
  * Hybrid repair (iliac artery stenting and common femoral artery reconstruction)
  * Endovascular repair (bare metal stenting, using covered stents, and plain balloon angioplasty)
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Short-term (30-days), mid-term (between 1-5 years), long-term (more than 5 years)
  Overall mortality in all treatment arms
Major adverse limb event (MALE) | Short-term (30-days), mid-term (between 1-5 years), long-term (more than 5 years)
  Major amputations (below and above the knee), new onset acute limb ischaemia of the treated extremity, and reintervention on the already treated arterial segment (aortoiliac segment and femoral bifurcation, excluding distal infrainguinal disease).

SECONDARY OUTCOMES:
30-day complication | Short-term (30-days)
  Major adverse cardiovascular events (MACE): myocardial infarction, heart failure, stroke, pulmonary embolism; acute kidney injury according to the RIFLE criteria (more than 50% increase of creatinine, and more than 50% drop of estimated glomerular filtration rate (eGFR) compared to the baseline preoperative values) three grades: Injury, Failure, Loss; blood transfusion, bowel ischaemia, urgent reintervention, thrombosis requiring reintervention, bleeding requiring reintervention, wound infection
Primary patency | Short-term (30-days), mid-term (between 1-5 years), long-term (more than 5 years)
  Computerized tomography or Doppler ultrasound findings of stenosis or occlusion (>50% stenosis defined as a >100% increase in the peak systolic velocity relative to the adjacent segments), or a combination of these findings

CONTACTS AND LOCATIONS:
Overall Officials: Joao Rocha Neves, MD PhD, Study Director — Univeristy of Porto
Locations (1):
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided
after the kick-up meeting we will ask all participating centres about their opinion on this decision, and at that moment final decision will be made

REFERENCES:
- [Result] Antonello M, Squizzato F, Bassini S, Porcellato L, Grego F, Piazza M. Open repair versus endovascular treatment of complex aortoiliac lesions in low risk patients. J Vasc Surg. 2019 Oct;70(4):1155-1165.e1. doi: 10.1016/j.jvs.2018.12.030. Epub 2019 Mar 6. PMID 30850298
- [Result] Mayor J, Branco BC, Chung J, Montero-Baker MF, Kougias P, Mills JL Sr, Gilani R. Outcome Comparison between Open and Endovascular Management of TASC II D Aortoiliac Occlusive Disease. Ann Vasc Surg. 2019 Nov;61:65-71.e3. doi: 10.1016/j.avsg.2019.06.005. Epub 2019 Aug 6. PMID 31394230
- [Result] Starodubtsev V, Mitrofanov V, Ignatenko P, Gostev A, Preece R, Rabtsun A, Saaya S, Popova I, Karpenko A. Editor's Choice - Hybrid vs. Open Surgical Reconstruction for Iliofemoral Occlusive Disease: A Prospective Randomised Trial. Eur J Vasc Endovasc Surg. 2022 Apr;63(4):557-565. doi: 10.1016/j.ejvs.2022.02.002. Epub 2022 Feb 9. PMID 35283003
- [Result] Suzuki K, Mizutani Y, Soga Y, Iida O, Kawasaki D, Yamauchi Y, Hirano K, Koshida R, Kamoi D, Tazaki J, Higashitani M, Shintani Y, Yamaoka T, Okazaki S, Suematsu N, Tsuchiya T, Miyashita Y, Shinozaki N, Takahashi H, Inoue N. Efficacy and Safety of Endovascular Therapy for Aortoiliac TASC D Lesions. Angiology. 2017 Jan;68(1):67-73. doi: 10.1177/0003319716638005. Epub 2016 Mar 15. PMID 26980775
- [Result] Squizzato F, D'Oria M, Bozza R, Porcellato L, Grego F, Lepidi S. Propensity-Matched Comparison of Endovascular versus Open Reconstruction for TASC-II C/D AortoIliac Occlusive Disease. A Ten-Year Single-Center Experience with Self-Expanding Covered Stents. Ann Vasc Surg. 2021 Feb;71:84-95. doi: 10.1016/j.avsg.2020.08.139. Epub 2020 Sep 11. PMID 32927036